CLINICAL TRIAL: NCT06256185
Title: Machine Learning to Predict Lymph Node Metastasis in T1 Esophageal Squamous Cell Carcinoma: A Multicenter Study
Brief Title: Machine Learning to Predict Lymph Node Metastasis in T1 Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 81902396
Record Dates: First submitted 2024-01-23; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Lymph Node Metastasis
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Esophagectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm used for predicting lymph node metastasis (Experimental)
  Interventions: Procedure: esophagectomy

INTERVENTIONS:
Procedure: esophagectomy — Resection of esophageal tumor and lymph node dissection

SUMMARY:
Existing models do poorly when it comes to quantifying the risk of Lymph node metastases (LNM). This study generated elastic net regression (ELR), random forest (RF), extreme gradient boosting (XGB), and a combined (ensemble) model of these for LNM in patients with T1 esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Lymph node metastases (LNM) is a relatively uncommon but possible complication of T1 esophageal squamous cell carcinoma (ESCC). Existing models do poorly when it comes to quantifying this risk. This study aimed to develop a machine learning model for LNM in patients with T1 esophageal squamous cell carcinoma.

Patients with T1 squamous cell carcinoma treated with surgery between January 2010 and September 2021 from 3 institutions were included in this study. Machine-learning models were developed using data on patients' age and sex, depth of tumor invasion, tumor size, tumor location, macroscopic tumor type, lymphatic and vascular invasion, and histologic grade. Elastic net regression (ELR), random forest (RF), extreme gradient boosting (XGB), and a combined (ensemble) model of these was generated. Use Area Under Curve (AUC) to evaluate the predictive ability of the model. The contribution to the model of each factor was calculated. In order to better meet clinical needs, the investigators have designed the model as a user-friendly website.

ELIGIBILITY:
Inclusion Criteria:

* (I) thoracic ESCC
* (II) no history of concomitant or prior malignancy
* (III) tumor with pT1 staging
* (IV) 15 or more lymph nodes examined

Exclusion Criteria:

* underwent neoadjuvant treatment or endoscopic submucosal dissection before surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1267 (Actual)
Dates: Start 2010-01-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Model performance: discrimination | 8 weeks
  Draw the ROC curve of the model and obtain their AUC values, and select the best prediction model based on the results of the validation set
Variable importance | 6 weeks
  Calculate the importance level of variables used in the model and sort them, and analyze the reasons for the most important variables
Sub-analysis (ML Model vs. Logistic Model vs. NCCN Guideline) | 8 weeks
  Apply NCCN guidelines and logistic models for prediction, and compare their performance with the model obtained in this study to determine the actual application benefits of the model

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erratum: Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2020 Jul;70(4):313. doi: 10.3322/caac.21609. Epub 2020 Apr 6. No abstract available. PMID 32767693
- [Background] Ohashi S, Miyamoto S, Kikuchi O, Goto T, Amanuma Y, Muto M. Recent Advances From Basic and Clinical Studies of Esophageal Squamous Cell Carcinoma. Gastroenterology. 2015 Dec;149(7):1700-15. doi: 10.1053/j.gastro.2015.08.054. Epub 2015 Sep 12. PMID 26376349
- [Background] Merkow RP, Bilimoria KY, Keswani RN, Chung J, Sherman KL, Knab LM, Posner MC, Bentrem DJ. Treatment trends, risk of lymph node metastasis, and outcomes for localized esophageal cancer. J Natl Cancer Inst. 2014 Jul 16;106(7):dju133. doi: 10.1093/jnci/dju133. Print 2014 Jul. PMID 25031273
- [Background] Alvarez Herrero L, Pouw RE, van Vilsteren FG, ten Kate FJ, Visser M, van Berge Henegouwen MI, Weusten BL, Bergman JJ. Risk of lymph node metastasis associated with deeper invasion by early adenocarcinoma of the esophagus and cardia: study based on endoscopic resection specimens. Endoscopy. 2010 Dec;42(12):1030-6. doi: 10.1055/s-0030-1255858. Epub 2010 Oct 19. PMID 20960392
- [Background] Gamboa AM, Kim S, Force SD, Staley CA, Woods KE, Kooby DA, Maithel SK, Luke JA, Shaffer KM, Dacha S, Saba NF, Keilin SA, Cai Q, El-Rayes BF, Chen Z, Willingham FF. Treatment allocation in patients with early-stage esophageal adenocarcinoma: Prevalence and predictors of lymph node involvement. Cancer. 2016 Jul 15;122(14):2150-7. doi: 10.1002/cncr.30040. Epub 2016 May 3. PMID 27142247
- [Background] Dubecz A, Kern M, Solymosi N, Schweigert M, Stein HJ. Predictors of Lymph Node Metastasis in Surgically Resected T1 Esophageal Cancer. Ann Thorac Surg. 2015 Jun;99(6):1879-85; discussion 1886. doi: 10.1016/j.athoracsur.2015.02.112. Epub 2015 Apr 28. PMID 25929888
- [Background] Zheng H, Tang H, Wang H, Fang Y, Shen Y, Feng M, Xu S, Fan H, Ge D, Wang Q, Tan L. Nomogram to predict lymph node metastasis in patients with early oesophageal squamous cell carcinoma. Br J Surg. 2018 Oct;105(11):1464-1470. doi: 10.1002/bjs.10882. Epub 2018 Jun 4. PMID 29863776
- [Background] Duan X, Shang X, Yue J, Ma Z, Chen C, Tang P, Jiang H, Yu Z. A nomogram to predict lymph node metastasis risk for early esophageal squamous cell carcinoma. BMC Cancer. 2021 Apr 20;21(1):431. doi: 10.1186/s12885-021-08077-z. PMID 33879102
- [Background] Collins GS, Dhiman P, Andaur Navarro CL, Ma J, Hooft L, Reitsma JB, Logullo P, Beam AL, Peng L, Van Calster B, van Smeden M, Riley RD, Moons KG. Protocol for development of a reporting guideline (TRIPOD-AI) and risk of bias tool (PROBAST-AI) for diagnostic and prognostic prediction model studies based on artificial intelligence. BMJ Open. 2021 Jul 9;11(7):e048008. doi: 10.1136/bmjopen-2020-048008. PMID 34244270
- [Background] Jiang KY, Huang H, Chen WY, Yan HJ, Wei ZT, Wang XW, Li HX, Zheng XY, Tian D. Risk factors for lymph node metastasis in T1 esophageal squamous cell carcinoma: A systematic review and meta-analysis. World J Gastroenterol. 2021 Feb 28;27(8):737-750. doi: 10.3748/wjg.v27.i8.737. PMID 33716451
- [Background] Pavlou M, Ambler G, Seaman SR, Guttmann O, Elliott P, King M, Omar RZ. How to develop a more accurate risk prediction model when there are few events. BMJ. 2015 Aug 11;351:h3868. doi: 10.1136/bmj.h3868. PMID 26264962
- [Background] van Vliet EP, Heijenbrok-Kal MH, Hunink MG, Kuipers EJ, Siersema PD. Staging investigations for oesophageal cancer: a meta-analysis. Br J Cancer. 2008 Feb 12;98(3):547-57. doi: 10.1038/sj.bjc.6604200. Epub 2008 Jan 22. PMID 18212745
- [Background] Choi J, Kim SG, Kim JS, Jung HC, Song IS. Comparison of endoscopic ultrasonography (EUS), positron emission tomography (PET), and computed tomography (CT) in the preoperative locoregional staging of resectable esophageal cancer. Surg Endosc. 2010 Jun;24(6):1380-6. doi: 10.1007/s00464-009-0783-x. Epub 2009 Dec 24. PMID 20033712
- [Background] Ou J, Wu L, Li R, Wu CQ, Liu J, Chen TW, Zhang XM, Tang S, Wu YP, Yang LQ, Tan BG, Lu FL. CT radiomics features to predict lymph node metastasis in advanced esophageal squamous cell carcinoma and to discriminate between regional and non-regional lymph node metastasis: a case control study. Quant Imaging Med Surg. 2021 Feb;11(2):628-640. doi: 10.21037/qims-20-241. PMID 33532263
- [Background] Wang S, Chen X, Fan J, Lu L. Prognostic Significance of Lymphovascular Invasion for Thoracic Esophageal Squamous Cell Carcinoma. Ann Surg Oncol. 2016 Nov;23(12):4101-4109. doi: 10.1245/s10434-016-5416-8. Epub 2016 Jul 19. PMID 27436201
- [Background] Li B, Chen H, Xiang J, Zhang Y, Kong Y, Garfield DH, Li H. Prevalence of lymph node metastases in superficial esophageal squamous cell carcinoma. J Thorac Cardiovasc Surg. 2013 Nov;146(5):1198-203. doi: 10.1016/j.jtcvs.2013.07.006. Epub 2013 Aug 26. PMID 23988285
- [Background] Shen W, Shen Y, Tan L, Jin C, Xi Y. A nomogram for predicting lymph node metastasis in surgically resected T1 esophageal squamous cell carcinoma. J Thorac Dis. 2018 Jul;10(7):4178-4185. doi: 10.21037/jtd.2018.06.51. PMID 30174862
- [Background] Akutsu Y, Uesato M, Shuto K, Kono T, Hoshino I, Horibe D, Sazuka T, Takeshita N, Maruyama T, Isozaki Y, Akanuma N, Matsubara H. The overall prevalence of metastasis in T1 esophageal squamous cell carcinoma: a retrospective analysis of 295 patients. Ann Surg. 2013 Jun;257(6):1032-8. doi: 10.1097/SLA.0b013e31827017fc. PMID 23108117
- [Background] Emi M, Hihara J, Hamai Y, Furukawa T, Ibuki Y, Okada M. Clinicopathologic Features of Submucosal Esophageal Squamous Cell Carcinoma. Ann Thorac Surg. 2017 Dec;104(6):1858-1864. doi: 10.1016/j.athoracsur.2017.06.037. Epub 2017 Oct 21. PMID 29033014

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT06256185/SAP_000.pdf